Title: TMS Alteration of the Reward Positivity

NCT05443256

Document Date: 02/24/2022

## **Statistical Analysis Plan**

Mean activity will be contrasted within-subjects as the subtraction of the stimulation condition from the sham condition. Given the small sample size of this pilot study, there are no plans to initiate frequentist statistical tests.